CLINICAL TRIAL: NCT04626778
Title: Clinical Efficacy of Single-Use of Peroxyl Mouthwash for Reducing Bacteria in Saliva and Bioaerosol Contamination Phase I
Brief Title: Clinical Efficacy of Single-Use of Peroxyl Mouthwash for Reducing Bacteria in Saliva and Bioaerosol Contamination
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Colgate Palmolive (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CRO-2020-08-BAC-HP-CA-BGS
Record Dates: First submitted 2020-11-05; First posted 2020-11-13 (Actual); Last update posted 2021-01-20 (Actual); Status verified 2020-11

CONDITIONS: Healthy
Keywords: Mouthwash; Saliva; Bioaerosol; Bacteria; Gingivitis
MeSH Terms: conditions — Gingivitis

STUDY DESIGN:
Intervention Model Description: Each subject will be randomized to receive one of the two possible study products.
Who Masked: Participant, Investigator
Masking Description: A blinded randomized controlled parallel group design trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Peroxyl (Active Comparator): 1.5% Hydrogen Peroxide mouthwash
  Interventions: Drug: Peroxyl Mouthwash
- placebo mouthwash (Placebo Comparator): 0.0% Hydrogen peroxide mouthwash
  Interventions: Drug: Placebo Mouthwash

INTERVENTIONS:
Drug: Peroxyl Mouthwash — Mouthwash
  Other Names: 1.5% HP
  Arms: Peroxyl
Drug: Placebo Mouthwash — Mouthwash
  Other Names: 0.0% HP Mouthwash
  Arms: placebo mouthwash

SUMMARY:
To evaluate the anti-bacterial, pre-procedural, clinical efficacy of Peroxyl mouthwash (1.5% hydrogen peroxide) in saliva and the reduction of bioaerosol contamination as compared to a matching placebo mouthwash (0.0% hydrogen peroxide)

DETAILED DESCRIPTION:
Qualified subjects will be enrolled and randomized to either one of the two study groups, balanced on the basis of their initial gingival index scores. Saliva samples will be collected from participants prior to rinsing with their assigned mouthwash (1.5% hydrogen peroxide or 0.0% hydrogen peroxide) for one minute and then expectorate. Saliva samples will again be collected immediately after, at 30 min, and 60 min after rinsing. All collected saliva samples will be placed in sterile vials, labeled with subject information and transferred to the microbiology laboratory for analysis.

ELIGIBILITY:
Inclusion Criteria:

* Potential subjects must meet ALL of the following criteria:

  * Subjects, ages 18-70, inclusive.
  * Availability for the duration of this clinical research study.
  * Good general health.
  * At least 20 natural teeth.
  * Gingivitis Index 1.0 (Löe-Silness).
  * Signed Informed Consent Form

Exclusion Criteria:

* Potential subjects must NOT HAVE ANY of the following conditions:

  * Symptoms consistent with COVID-19 or have tested positive.
  * Presence of orthodontic bands.
  * Tumor(s) of the soft or hard tissues of the oral cavity.
  * Advanced periodontal disease (purulent exudate, tooth mobility, and/or extensive loss of periodontal attachment or alveolar bone) or peri-implantitis.
  * Five or more carious lesions requiring immediate restorative treatment.
  * Use of antibiotic one-month prior to entry into the study.
  * Participation in any other clinical study or test panel within the one month prior to entry into the study.
  * Dental prophylaxis during the past two weeks prior to baseline examinations.
  * History of allergies to oral care/personal care consumer products or their ingredients.
  * On any prescription medicines that might interfere with the study outcome.
  * An existing medical condition that prohibits not eating or drinking for periods up to 4 hours.
  * History of alcohol or drug abuse.
  * Self-reported pregnant or lactating subjects.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2020-10-08 (Actual); Primary Completion 2020-12-15 (Actual); Study Completion 2020-12-15 (Actual)

PRIMARY OUTCOMES:
Change in the Colony Forming Unit of total bacteria in saliva and in bioaerosol | baseline, 30 minutes & 60 minutes
  Saliva samples will be collected from participants prior to rinsing with their assigned mouthwash (1.5% hydrogen peroxide or 0.0% hydrogen peroxide) for one minute and then expectorate. Saliva samples will again be collected immediately after, at 30 min, and 60 min after rinsing. All collected saliva samples will be placed in sterile vials, labeled with subject information and transferred to the microbiology laboratory for analysis.

CONTACTS AND LOCATIONS:
Overall Officials: Yiming Li, DDS/PhD/MSD, Principal Investigator — Loma Linda University School of Dentistry, Center for Dental Research
Locations (1):
- Loma Linda University School of Dentistry, Center for Dental Research, Loma Linda, California, United States

IPD SHARING:
Plan to Share IPD: Yes
All IPD that underlie results in a publication
Supporting Information: Study Protocol
Time Frame: after analysis is completed